CLINICAL TRIAL: NCT05023590
Title: Monocentric, Randomized, Prospective Study to Compare Endocardiac Radio Frequency Ablation and Cryo Ablation of the Left Atrium During an Open Chest Mitral Valve Intervention
Brief Title: Atrial Fibrillation Registry 2017
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Herz- und Gefaesszentrum Bad Bevensen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHA17-Registry
Record Dates: First submitted 2021-05-05; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation; Mitral Valve Failure
Keywords: sinus rhythm; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: monocentric, 1:1 randomized (cryo ablation vs. radiofrequency ablation), open-label, parallel, registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryo ablation (Active Comparator): cryo ablation of left atrium during mitral valve open chest intervention
  Interventions: Procedure: ablation of left atrium during mitral valve open chest intervention
- radio frequency ablation (Active Comparator): radio frequency ablation of left atrium during mitral valve open chest intervention
  Interventions: Procedure: ablation of left atrium during mitral valve open chest intervention

INTERVENTIONS:
Procedure: ablation of left atrium during mitral valve open chest intervention — open chest mitral valve surgery (reconstruction or replacement) with additional ablation of left atrium by cryo or radio frequency method

SUMMARY:
Monocentric, prospective, randomized trial of cardiac surgical arrhythmia using endocardial radiofrequency atrial ablation compared with a cryo ablation system in the setting of cardiac surgery.

DETAILED DESCRIPTION:
Regular, rhythmic monitoring (24-hour Holter ECG, 5 and 28 days, 3 and 6 months po) of patients after cardiac surgery on the mitral valve with atrial ablation for paroxysmal, persistent, and permanent atrial fibrillation with regard to the presence or stability of sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Present, written informed consent from the patient
* paroxysmal, persistent, or permanent atrial fibrillation not longer than 10 years according to guidelines (ACC, AHA, ESC)
* planned cardiac surgery on the mitral valve
* ECHO parameters : LA size a.p. ≤ 55mm

Exclusion Criteria:

* permanent atrial fibrillation longer than 10 years
* ECHO parameters : LA size a.p. > 55mm
* pregnancy
* life expectancy < 12 months
* lack of cognitive or mental capacity to participate in the study
* Patients who are to be included in another clinical (interventional) study at the same time or who are already participating in such a study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
number of patients with stabil sinus rhythm 6 month after ablation | 6 month after index surgery / ablation
  number of patients with stabil sinus rhythm 6 month after ablation

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Wimmer-Greinecker, Prof., Principal Investigator — Herz- und Gefäßzentrum Bad Bevensen
Locations (1):
- Herz- und Gefaesszentrum Bad Bevensen, Bad Bevensen, Lower Saxony, Germany